CLINICAL TRIAL: NCT01749189
Title: A Randomized, Controlled Double Blind Longitudinal Study: Effect of Protein Blend Supplementation During Exercise Training on Muscle Growth and Strength
Brief Title: Effect of Protein Blend Supplementation During Exercise Training on Muscle Growth and Strength
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DuPont Nutrition and Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CRC-D-179
Record Dates: First submitted 2012-11-15; First posted 2012-12-13 (Estimated); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Muscle
Keywords: soy; whey; casein; muscle; strength; protein
MeSH Terms: interventions — Whey

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo dry blended beverage (carbohydrate)
  Interventions: Dietary Supplement: Placebo
- Blend (Experimental): A dry blended beverage containing a protein blend of soy, whey and casein
  Interventions: Dietary Supplement: Blend
- Whey (Active Comparator): A dry blended beverage containing Whey protein
  Interventions: Dietary Supplement: Whey

INTERVENTIONS:
Dietary Supplement: Blend — 22 grams of protein/day
  Arms: Blend
Dietary Supplement: Whey — 22 grams of protein/day
  Arms: Whey
Dietary Supplement: Placebo — 22 grams of carbohydrate/day
  Arms: Placebo

SUMMARY:
This study will investigate the effects of a soy/dairy protein blend on muscle growth and strength. In sports nutrition and in aging it is important to have healthy muscles. This can be achieved with exercise and nutrition. Consumption of protein following resistance exercise can promote healthy muscle growth and help improve strength. Young healthy men will be studied during a 12 week resistance exercise training program and be given protein supplements every day during the study. The hypothesis is that a blend of soy, whey and casein will induce a greater muscle gain and strength increase than the control.

ELIGIBILITY:
Inclusion Criteria:

* Stable body weight, healthy, males aged 18-35

Exclusion Criteria:

1. Exercise training (>2 weekly sessions of moderate to high intensity aerobic or resistance exercise)
2. Resistance Training (>2 weekly sessions of moderate to high intensity) within the past six months
3. Any orthopedic injury that prohibits participation in the exercise training
4. Significant heart, liver, kidney, blood, or respiratory disease
5. Peripheral vascular disease
6. Diabetes mellitus or other untreated endocrine disease
7. Active cancer (all groups) and history of cancer
8. Acute infectious disease or history of chronic infections (e.g. TB, hepatitis, HIV, herpes)
9. Recent (within 6 months) treatment with anabolic steroids, or corticosteroids.
10. Alcohol or drug abuse
11. Tobacco use (smoking or chewing)
12. BMI range will be (20-29.9 kg/m2) to exclude for Malnutrition (hypoalbuminemia, and/or hypotransferrinemia) and Obesity
13. Low hemoglobin levels (below normal values)
14. Food allergies (including milk and soy)
15. Individuals on a Vegetarian Diet
16. Females
17. Average protein intake < 0.6 or >1.8 g/kg per day
18. Taking dietary supplements such as green tea, creatine, ribose, whey or soy protein, etc. within the past 6 months
19. Currently on a high-soy diet or high dairy diet (consuming >2 servings of soy per day or >6 servings of dairy)

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2012-07; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change in Muscle Mass | Baseline, 6 weeks, 12 weeks
  Muscle Mass will be determined by DEXA

SECONDARY OUTCOMES:
Change in Muscle Strength | Baseline, 6 weeks, 12 weeks
  Knee Extensor

CONTACTS AND LOCATIONS:
Overall Officials: Blake Rasmussen, PhD, Principal Investigator — University of Texas; Mark B Cope, PhD, Principal Investigator — Solae, LLC
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

REFERENCES:
- [Derived] Reidy PT, Fry CS, Igbinigie S, Deer RR, Jennings K, Cope MB, Mukherjea R, Volpi E, Rasmussen BB. Protein Supplementation Does Not Affect Myogenic Adaptations to Resistance Training. Med Sci Sports Exerc. 2017 Jun;49(6):1197-1208. doi: 10.1249/MSS.0000000000001224. PMID 28346813
- [Derived] Reidy PT, Borack MS, Markofski MM, Dickinson JM, Deer RR, Husaini SH, Walker DK, Igbinigie S, Robertson SM, Cope MB, Mukherjea R, Hall-Porter JM, Jennings K, Volpi E, Rasmussen BB. Protein Supplementation Has Minimal Effects on Muscle Adaptations during Resistance Exercise Training in Young Men: A Double-Blind Randomized Clinical Trial. J Nutr. 2016 Sep;146(9):1660-9. doi: 10.3945/jn.116.231803. Epub 2016 Jul 27. PMID 27466602